CLINICAL TRIAL: NCT03671291
Title: National Survey on Missed Opportunities to Pre-exposure Prophylaxis for Prevention of Human Immunodeficiency Virus-infection.
Brief Title: Missed Opportunities to Pre-exposure Prophylaxis for HIV Infection on Person Newly Diagnosed With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: University Hospital, Marseille (Other); University Hospital, Grenoble (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Montpellier (Other); Hospital Purpan (Other); University Hospital, Bordeaux (Other); Hôpital de la Croix-Rousse (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital of Saint-Etienne (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire de Besancon (Other); Tourcoing Hospital (Other); University Hospital, Strasbourg (Other); Nantes University Hospital (Other); Centre Hospitalier Régional d'Orléans (Other); Rennes University Hospital (Other); Saint Antoine University Hospital (Other); Tenon Hospital, Paris (Other); Saint-Louis Hospital, Paris, France (Other); Hôpital Necker-Enfants Malades (Other); Bicetre Hospital (Other); Pitié-Salpêtrière Hospital (Other); Bichat Hospital (Other); University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 95041 Missed Opportunity
Record Dates: First submitted 2018-09-05; First posted 2018-09-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Virus-HIV
Keywords: VIH; PrEP; risk factors; Prevention; Access to care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recently infected with HIV (Experimental): Men and women recently infected with HIV and have been eligible for PrEP based on the recommendation of french national regulatory agency regarding the prescription of Truvada® in prophylaxis to HIV exposure. The potential reasons behind these missed opportunity of Pre-exposure prophylaxis will be studied through a self-administrated questionnaire.
  Interventions: Behavioral: self-administrated questionnaire

INTERVENTIONS:
Behavioral: self-administrated questionnaire — Persons who the biological parameters or past screening show that they were recently infected with HIV cf. eligibility criteria, will, after obtaining his consent, answer a series of questions through a self-administrated questionnaire that will take approximately 40 minutes.

SUMMARY:
Missed opportunity to pre-exposure prophylaxis is a survey study that will be addressed to newly infected with human immunodeficiency virus (HIV) persons. The purposes of this study is to understand why despite the fact that pre-exposure prophylaxis exist, these persons have been contaminated with HIV.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis is a new strategy to prevent the occurrence of new cases of HIV. This prophylaxis strategy is based on taking antiretroviral drugs (ARV) before and after exposition to a risk of HIV infection which can reduce drastically the contamination with HIV. A certain groups of population based on their sexual orientation, for instance man who have sex with man (MSM), is among the groups that are highly exposed to this risk. To reduce this risk, French national regulatory authority (ANSM), firstly through temporary usage recommendation followed by a marketing authorization extension, allowed the prescription of these antiretroviral molecules to persons presenting eligibility criteria as defined by regulatory authority. Despite these preventive measures, the incidence of HIV such as the MSM group still high. The missed opportunity studies has as objectives to try to disentangle real obstacles of PrEP use in France and to optimize PrEP criteria if needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Understanding and speaking French
* Affiliated in or beneficiary of a Social Security (excluding State Medical Aid or AME that aren't considered as Social Security coverage)
* Men and women with a diagnosis of HIV infection known for less than three months and with recent HIV infection established on:

a diagnostic confirmation test by Western Blot (WB) or Immuno Blot showing incomplete pattern.

OR Previous HIV negative screening test performed within 6 months of diagnosis.

Exclusion Criteria:

* Less than 18 years old
* Unable to understand French
* Not affiliated to a social security coverage
* Under guardianship or under curatorship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients eligible for PrEP at the time of HIV infection | The needed time to answer to the questionnaire : 40 min to 1 hour.
  Quantify and describe among newly diagnosed people with HIV the missed opportunities for PrEP treatment for HIV infection prevention

SECONDARY OUTCOMES:
Taking a risky behaviour for HIV infection | The needed time to answer to the questionnaire : 40 min to 1 hour.
  Better identify risk taking exposures to HIV contamination and determine the adequacy of the criteria for access to pre-exposure treatment with current practices. For this, questions concerning the frequency of unprotected sex, the number of partners and the type of sexual practices are collected in the self-questionnaire.
Awareness and level of knowledge of the PrEP strategy | The needed time to answer to the questionnaire : 40 min to 1 hour.
  Study the individual factors associated with the knowledge, representations, acceptance and prescription of PrEP in order to evaluate the hindrance to the establishment of PrEP and the persistence of infections despite the availability of this new strategy of preventive treatment. For this, the questionnaire asks about the knowledge of the existence of this prevention tool, the antecedent of PrEP intake, and the potential reasons for not taking PrEP.
Access to care | The needed time to answer to the questionnaire : 40 min to 1 hour.
  Evaluate the impact of healthcare professionals on missed opportunities for PrEP through the access to general or hospital physicians and screening history. Comparing percentage of new infections among new HIV diagnosis in order to study regional disparities in term of HIV screening access according to city/region and area.
  Access to care, meaning frequency of visit to, the nature of, health care facilities (hospital, urban doctor, anonymous screening center…), discussed items during consultation with physician etc. These kind of informations will help to appreciate if access to care in all its dimension is correlated to HIV infection risk.
  These different criteria will be compared by region to determine whether regional disparities in access to care occurred.
Availability of PrEP | The needed time to answer to the questionnaire : 40 min to 1 hour.
  Study the structural and demographic factors associated with missed opportunities for PrEP (regional disparities in access to PrEP).
  A questionnaire for each participating center asks about the type of consultations offered, the presence of specific consultations and support for PrEP, the active file of people under PrEP and will determine if there is a center and / or region effect for taking PrEP. Collected information will shed the light on potential relation between logistic means and availability of PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Poizot-Martin, Dr, Principal Investigator — Centre d'Informations et de soins de l'Immunodéficience Humaine et des hépatites Virales- CHU Sainte-Marguerite
Locations (1):
- Centre d'Informations et de soins de l'Immunodéficience Humaine et des hépatites Virales- CHU Sainte-Marguerite, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided
We need to make a concertation with PI and scientists.